CLINICAL TRIAL: NCT04713969
Title: Duodenal Neuro-immune Interactions and Effects of PPI in Functional Dyspepsia
Brief Title: Neuro-immune Interactions and PPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S64807/64847
Record Dates: First submitted 2020-12-17; First posted 2021-01-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-06

CONDITIONS: Functional Dyspepsia
Keywords: inflammation; imaging
MeSH Terms: conditions — Inflammation | interventions — Pantoprazole

STUDY DESIGN:
Intervention Model Description: Intervention with PPI (Pantoprazole 40mg twice daily) in 30 FD patients. Baseline procedures in 30 healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional dyspepsia patients before and after PPI (Experimental): Pantoprazole 40mg twice daily in functional dyspepsia patients for 4 weeks
  Interventions: Drug: Pantoprazole 40mg
- Healthy controls without PPI (No Intervention): Baseline investigations

INTERVENTIONS:
Drug: Pantoprazole 40mg — Pantoprazole 40mg twice daily
  Other Names: Pantomed
  Arms: Functional dyspepsia patients before and after PPI

SUMMARY:
Prospective interventional study on duodenal neuro-immune interactions in healthy volunteers and functional dyspepsia patients and the effects of PPI

DETAILED DESCRIPTION:
Duodenal low-grade inflammation is frequently reported in functional dyspepsia (FD), while also neuronal and structural changes in duodenal submucosal ganglia have been described in FD patients. Proton pump inhibitors (PPI) are the first-line therapy in FD patients and are recently shown to have anti-inflammatory properties in FD. However, the exact mechanism of their anti-inflammatory action is unknow and their effect on duodenal nerve signalling remain unclear.

In this prospective interventional study, FD patients will undergo study procedures before and after treatment with pantoprazole (Pantomed®) 40mg twice daily during 4 weeks, with a baseline comparison to healthy volunteers.

This study aims to provide an in-deep characterization of the inflammatory infiltrate in the duodenum of FD patients, and to unravel the effect of PPI-therapy on neuronal signalling, duodenal inflammation and neuro-immune interactions in FD.

Novel insights in the pathophysiology of FD, including the duodenal mucosal inflammation and impaired neuronal functioning, can provide a better understanding of this commonly and costly disorder. Moreover, these results will help to elucidate the anti-inflammatory effect of PPI, which will contribute to the discovery of predictive markers for therapeutic efficacy of PPI in FD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with FD diagnosis as per Rome IV criteria (EPS or PDS).
* Normal investigation including upper GI endoscopy.
* Patients have confirmed duodenal mucosal eosinophilia.
* Patients witnessed written informed consent.
* Patients aged between 18 and 64 years inclusive.
* Male or female (not pregnant or lactating and using contraception or postmenopausal).
* Subjects are capable to understand the study and the questionnaires, and to comply with the study requirements.

Exclusion Criteria:

* Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study.
* Patients with any major psychiatric disorders (stable dose of single antidepressant allowed for psychiatric indication, no limitation for other indications).
* Patients presenting with predominant symptoms of irritable bowel syndrome (IBS) or of gastro-esophageal reflux disease (GERD).
* Patients with personal or family (first-degree relative) of diabetes mellitus, celiac disease, inflammatory bowel disease, psoriasis, lupus, scleroderma, rheumatic or other systemic auto-immune disease.
* Patients with eosinophilic esophagitis or eosinophilic gastroenteritis.
* Active H. pylori infection (or <6 months after eradication).
* Allergy or atopy, including therapy.
* Organic gastro-intestinal disease or history of gastrointestinal surgery other than appendectomy or splenectomy.
* Known impaired liver or kidney dysfunction, or coagulation disorders.
* Known HIV, HBV or HCV infection, including therapy.
* Active coronary or peripheral artery disease.
* Use of anti-inflammatory drugs or anti-allergy drugs <2 weeks before sampling.
* Use of immunosuppressants, antibiotics or acid-suppressive drugs <3 months before sampling.
* Use of prokinetics <2 weeks before sampling (unless if ≤3/week).
* Significant alcohol use (>10 units/week).
* Any use of alcohol or smoking <2 days before sampling.
* Active malignancy, including therapy.
* Females who are pregnant or lactating.
* Patients not capable to understand or be compliant with the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
The effect of PPI on duodenal mucosal inflammation (assessed by flow cytometry on lamina propria leukocytes) in FD | 4 weeks
  Duodenal mucosal inflammation as assessed by flow cytometric quantification of immune cell populations in isolated lamina propria leukocytes before and after PPI

SECONDARY OUTCOMES:
The effect of PPI on symptoms (Patient Assessment of Upper Gastrointestinal Disorders - Symptom severity index [PAGI-SYM]) in FD | 4 weeks
  PAGI-SYM symptom scores (ranging from 0 [no symptoms] to 5 [very severe symptoms]) before and after PPI
The effect of PPI on quality of life (Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life [PAGI-QOL]) in FD | 4 weeks
  PAGI-QOL scores (ranging from 0 [lowest quality of life] to 5 [highest quality of life]) before and after PPI
The effect of PPI on salivary cortisol in FD | 4 weeks
  salivary cortisol before and after PPI
The effect of PPI on systemic inflammation (assessed by flow cytometry) in FD | 4 weeks
  Systemic inflammation quantified by flow cytometry of peripheral blood leukocytes before and after PPI

OTHER OUTCOMES:
The effect of PPI on calcium transient amplitudes after electrical stimulation of submucosal neurons in FD | 4 weeks
  Calcium transient amplitudes after electrical stimulation of interconnecting fiber bundles before and after PPI
The effect of PPI on urine metabolites in FD | 4 weeks
  urine metabolites before and after PPI

CONTACTS AND LOCATIONS:
Overall Officials: Tim Vanuytsel, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgie, Belgium

IPD SHARING:
Plan to Share IPD: No